CLINICAL TRIAL: NCT05064878
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Fixed-Dose, Multicenter Study To Examine The Efficacy And Safety Of ZX008 In Subjects With CDKL5 Deficiency Disorder Followed By An Open-Label Extension
Brief Title: A Study to Investigate the Efficacy and Safety of ZX008 in Subjects With CDKL5 Deficiency Disorder
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZX008-2103/EP0216; 2021-003222-76 (EudraCT Number); U1111-1303-2043 (Other: WHO universal trial number (UTN))
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: CDKL5 Deficiency Disorder; Generalized Tonic Clonic Seizure; Epileptic Spasm; Refractory Seizures
MeSH Terms: conditions — CDKL5 deficiency disorder; Epilepsy, Tonic-Clonic; Spasms, Infantile; Seizures | interventions — Fenfluramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ZX008 0.8 mg/kg/day (Experimental): Part 1: ZX008 0.8 mg/kg/day will be administered twice a day (BID) in equally divided doses; maximum of 30 mg/day, (subjects taking concomitant stiripentol will receive 0.5 mg/kg/day, [maximum of 20 mg/day]) with or without food.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)
- Placebo (Placebo Comparator): Part 1: Matching ZX008 placebo will be administered twice a day (BID) in equally divided doses with or without food.
  Interventions: Drug: Matching ZX008 Placebo
- ZX008 (Experimental): Part 2: Open-label ZX008 will be administered using a flexible dosing regimen, up to ZX008 0.8 mg/kg/day; maximum dose: 30 mg/day (subjects taking concomitant stiripentol will receive 0.5 mg/kg/day, [maximum of 20 mg/day]). ZX008 will be administered twice a day (BID) in equally divided doses with or without food.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride) — ZX008 is supplied as an oral aqueous solution of Fenfluramine Hydrochloride.
  Arms: ZX008; ZX008 0.8 mg/kg/day
Drug: Matching ZX008 Placebo — Matching ZX008 placebo is supplied as an oral solution.
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, parallel-group, placebo controlled, 2-part study to evaluate the efficacy and safety of ZX008 when used as adjunctive therapy for the treatment of uncontrolled seizures in children and adults with cyclin-dependent kinase like-5 (CDKL5) deficiency disorder (CDD).

DETAILED DESCRIPTION:
This is a 2-part multicenter trial. Part 1 is a 20-week randomized, double-blind, placebo-controlled, fixed-dose, parallel-group study to examine the efficacy and safety of ZX008 as an adjunctive therapy (to existing concomitant treatment with antiepileptic treatments [AETs]) in children and adults with a CDD diagnosis and uncontrolled seizures.

Part 1 of the study is 20 weeks in duration and will consist of the following stages: Baseline Period (ie, Baseline [BL]; 4 weeks including the Screening Visit and baseline observation), Titration Period (ie, Titration; 2 weeks), Maintenance Period (ie, Maintenance; 12 weeks), and a 2-week Transition Period (ie, Transition; 2 weeks) to the open-label starting dose.

Part 2 is a 54-week, open-label, flexible-dose, long-term extension for subjects who complete Part 1. Part 2 includes an Open-Label Extension (OLE) Treatment Period (52 weeks) with a Taper Period (ie, Taper; 2 weeks).

The primary study analysis to evaluate the efficacy and safety of ZX008 in children and adults with CDD will be based on Part 1 data in all randomized subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed pathogenic or likely pathogenic mutation in the CDKL5 gene and a clinical diagnosis of CDD with epilepsy onset in the first year of life, plus motor and developmental delays.
* Subject is male or female, aged 1 to 35 years, inclusive, as of the day of the Screening Visit.
* Subject must have failed to achieve seizure control despite previous or current use of 2 or more AETs.
* Subject is currently receiving at least 1 concomitant antiseizure treatment: antiseizure medication (ASM), vagus nerve stimulation (VNS), responsive neurostimulation (RNS), or ketogenic diet (KD).
* All medications or interventions for epilepsy (including VNS, RNS, and KD) must be stable prior to screening and are expected to remain stable throughout the study.
* At the Screening Visit, parent/caregiver reports that subject has ≥ 4 countable motor seizures(CMS) per week.

Exclusion Criteria:

* Subject has a known hypersensitivity to fenfluramine or any of the excipients in the study drug.
* Subject has a diagnosis of pulmonary arterial hypertension.
* Subject has a clinically significant medical condition, including chronic obstructive pulmonary disease, interstitial lung disease, or portal hypertension, or has had clinically relevant symptoms or a clinically significant illness currently or in the 4 weeks prior to the Screening Visit, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.
* Subject has current or past history of cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction or stroke, severe ventricular arrhythmias, or clinically significant structural cardiac abnormality, including but not limited to mitral valve prolapse, atrial or ventricular septal defects, patent ductus arteriosus, and patent foramen ovale with reversal of shunt. (Note: Patent foramen ovale or a bicuspid aortic valve are not considered exclusionary).
* Subject has moderate to severe hepatic impairment.
* Subject has current eating disorder that suggests anorexia nervosa or bulimia.
* Subject has a current or past history of glaucoma.
* Subject is taking > 4 concomitant ASMs. Rescue medications are not included in the count.
* Subject is receiving concomitant treatment with cannabidiol (CBD) other than Epidiolex/Epidyolex or is being actively treated with tetrahydrocannabinol (THC) or any marijuana product for any condition.
* Subject has participated in another interventional clinical trial within 30 days of the Screening Visit or is currently receiving an investigational product.
* Subject has previously been treated with Fintepla® (fenfluramine) prior to the Screening Visit.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2027-11-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
The median percentage change from the Baseline Period (Baseline) in "monthly (28 days) countable motor seizure frequency | 14 Weeks
  The median percentage change from the Baseline Period (Baseline) in "monthly (28 days) countable motor seizure frequency," or CMSF, during the combined Titration and Maintenance Periods (T+M) in the ZX008 0.8 mg/kg/day group compared with the placebo group

SECONDARY OUTCOMES:
The percentage of subjects who achieve a ≥ 50% reduction from Baseline in CMSF | 14 Weeks
  The percentage of subjects who achieve a ≥ 50% reduction from Baseline in CMSF during T+M in the ZX008 0.8 mg/kg/day group compared with the placebo group
The percentage of subjects who achieve improvement in the Clinical Global Impression-Improvement (CGI-I) rating as assessed by the Investigator | 14 Weeks
  The percentage of subjects who achieve a CGI-I rating of much or very much improved as assessed by the Investigator at the end of T+M in the ZX008 0.8 mg/kg group compared with the placebo group
The median percentage change from Baseline in monthly Generalized Tonic-Clonic (GTC) seizure frequency | 14 Weeks
  The median percentage change from Baseline in monthly GTC seizure frequency during T+M in the ZX008 0.8 mg/kg/day group compared with the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (46):
- United States (13):
  - Ep0216 154, Birmingham, Alabama
  - Ep0216 144, Los Angeles, California
  - Ep0216 101, San Francisco, California
  - Ep0216 173, Aurora, Colorado
  - Ep0216 149, Washington D.C., District of Columbia
  - Ep0216 157, Atlanta, Georgia
  - Ep0216 113, Boston, Massachusetts
  - Ep0216 134, Detroit, Michigan
  - Ep0216 166, Chapel Hill, North Carolina
  - Ep0216 164, Cleveland, Ohio
  - Ep0216 120, Philadelphia, Pennsylvania
  - Ep0216 124, Memphis, Tennessee
  - Ep0216 171, Austin, Texas
- Ep0216 2505, Linz, Austria
- Belgium (2):
  - Ep0216 804, Brussels
  - Ep0216 801, Edegem
- Ep0216 2802, Tbilisi, Georgia
- Germany (4):
  - Ep0216 902, Bielefeld
  - Ep0216 909, Kehl-Kork
  - Ep0216 908, Kiel
  - Ep0216 901, Vogtareuth
- Ep0216 1803, Dublin, Ireland
- Israel (3):
  - Ep0216 1909, Petah Tikva
  - Ep0216 1906, Ramat Gan
  - Ep0216 1904, Tel Aviv
- Italy (6):
  - Ep0216 1201, Florence
  - Ep0216 1204, Genova
  - Ep0216 1212, Modena
  - Ep0216 1206, Roma
  - Ep0216 1208, Roma
  - Ep0216 1202, Verona
- Japan (4):
  - Ep0216 1512, Hiroshima
  - Ep0216 1505, Niigata
  - Ep0216 1518, Ōmura
  - Ep0216 1502, Shizuoka
- Ep0216 1401, Zwolle, Netherlands
- Portugal (2):
  - Ep0216 2104, Lisbon
  - Ep0216 2105, Porto
- Spain (3):
  - Ep0216 1103, Barcelona
  - Ep0216 1117, Madrid
  - Ep0216 1118, Santiago de Compostela
- Ep0216 3101, Dubai, United Arab Emirates
- United Kingdom (4):
  - Ep0216 607, Bristol
  - Ep0216 602, London
  - Ep0216 611, Manchester
  - Ep0216 604, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org